CLINICAL TRIAL: NCT00234364
Title: Pergolide Treatment and Valvular Heart Disease
Status: Completed | Type: Observational
Sponsor: Århus Amt (Other Government)
Other Study IDs: permax
Record Dates: First submitted 2005-10-04; First posted 2005-10-07 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Heart Valve Diseases; Parkinson's Disease; Pergolide; Fibrosis
Keywords: Pergolide; Ergotamine derivates; Valvular heart disease
MeSH Terms: conditions — Heart Valve Diseases; Parkinson Disease; Fibrosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
In a blinded echocardiographic study we investigate the frequency of valvular abnormalities in a group of Parkinson patients treated with either ergot derived dopamine agonists (pergolide and cabergoline) or non-ergot derived dopamine agonists (pramipexole and ropinirole). The ability to detect patients with valvular abnormalities by clinical approach is examined.

DETAILED DESCRIPTION:
Some case reports and a single study, which included 78 Parkinson patients, has found a correlation between treatment with the ergotamine derivative dopamine agonists (pergolide) and restrictive valvular heart disease. The mechanisms are thought to be the same as with the former used anorectikum, fenfluramine and other drugs stimulating the 5HT-2B receptor.

In a blinded manner we make physiologic and echocardiographic examination on 160 Parkinson patients treated with either ergotamine or non-ergotamine derivative dopamine agonists (80 patients in each group) to see whether Parkinson patients treated with ergotamine derivatives have more heart valvular disease

ELIGIBILITY:
Inclusion Criteria:

* Parkinson patients who in the last year has been treated minimum 6 months with either ergotamine derivative or non-ergotamine derivative dopamine agonists (the latter included as controls)
* Informed contests

Exclusion Criteria:

* Control patients will be excluded if the have been treated with ergotamine derivates in the last 12 months or if the prior to that have had ergotamine derivates for more than 6 months
* Patients with known valvular heart disease prior to the diagnosis of Parkinson

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2005-03; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke G Rasmussen, MD, Principal Investigator — Aarhus University Hospital Skejby
Locations (1):
- Skejby Hospital, Aarhus, Aahus N, Denmark